CLINICAL TRIAL: NCT00057577
Title: Prevention of Recurrence in Depression With Drugs and CT
Acronym: CPT3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Steven Hollon, Professor of Psychology, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01MH060713 (NIH); R01MH060713 (NIH)
Record Dates: First submitted 2003-04-04; First posted 2003-04-07 (Estimated); Results first posted 2015-04-02 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Cognitive Behavioral Therapy; Dosage Forms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive therapy plus medications (Experimental): Participants will receive antidepressant medication plus cognitive therapy
  Interventions: Behavioral: Cognitive Therapy; Drug: Medications
- Medications alone (Experimental): Participants will receive maintenance of antidepressant medication alone
  Interventions: Drug: Medications

INTERVENTIONS:
Behavioral: Cognitive Therapy — CT sessions occur weekly during acute treatment and monthly during continuation. Acute treatment may last up to 18 months. Remitted patients are continued on medication for up to 36 months from initial randomization until they meet criteria for recovery. At recovery, patients receiving combined treatment discontinue CT.
  Other Names: CT
  Arms: Cognitive therapy plus medications
Drug: Medications — Antidepressant medication is distributed as clinically indicated with augmentation and ancillary medications as needed. Acute treatment may last up to 18 months. Remitted patients are continued on medication for up to 36 months from the point of initial randomization until they meet criteria for recovery. All recovered patients are randomized a second time to either maintenance medication or medication withdrawal. Patients are then monitored over 36 months to ascertain risk for recurrence of depressive symptoms.
  Other Names: ADM

SUMMARY:
This study will determine whether the addition of Cognitive Therapy (CT) to antidepressant medication (ADM) enhances treatment for depression. This study will also test whether the addition of CT to ADM will prevent recurrences of depression after therapy is over.

DETAILED DESCRIPTION:
It is commonly believed that the combination of ADM and psychotherapy is more effective in treating depression than either treatment alone. Data indicate that CT enhances the initial effects of ADM, but little research has been conducted to determine whether prior exposure to CT prevents the onset of new depressive episodes. This study will determine the effectiveness of adding CT to ADM for the treatment of depression.

Participants are randomly assigned to receive either ADM alone or ADM plus CT for up to 18 months. Remitted patients are continued on medication for up to 36 months from the point of initial randomization until they meet criteria for recovery. At recovery, patients receiving combined treatment discontinue cognitive therapy; all recovered patients are randomized a second time to either maintenance medication or medication withdrawal. Patients are then monitored over 36 months to ascertain risk for recurrence of depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent or chronic major depressive disorder

Exclusion Criteria:

* Current diagnosis of psychotic affective disorder
* History of nonaffective psychotic disorder
* Substance dependence last three months requiring detox
* Schizotypal, antisocial, or borderline personality disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2002-10; Primary Completion 2012-07 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven D. Hollon, PhD, Principal Investigator — Vanderbilt University; Robert J. DeRubeis, PhD, Principal Investigator — University of Pennsylvania; Jan A. Fawcett, MD, Principal Investigator — Rush Medical Center
Locations (3):
- United States (3):
  - Rush Medical Center - Treatment Research Unit, Chicago, Illinois
  - Depression Research Unit, University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt Adult Outpatient Psychiatry, Nashville, Tennessee

REFERENCES:
- [Derived] Khazanov GK, Xu C, Hollon SD, DeRubeis RJ, Thase ME. Adding cognitive therapy to antidepressant medications decreases suicidal ideation. J Affect Disord. 2021 Feb 15;281:183-191. doi: 10.1016/j.jad.2020.12.032. Epub 2020 Dec 8. PMID 33326891
- [Derived] Khazanov GK, Xu C, Dunn BD, Cohen ZD, DeRubeis RJ, Hollon SD. Distress and anhedonia as predictors of depression treatment outcome: A secondary analysis of a randomized clinical trial. Behav Res Ther. 2020 Feb;125:103507. doi: 10.1016/j.brat.2019.103507. Epub 2019 Oct 31. PMID 31896529
- [Derived] DeRubeis RJ, Zajecka J, Shelton RC, Amsterdam JD, Fawcett J, Xu C, Young PR, Gallop R, Hollon SD. Prevention of Recurrence After Recovery From a Major Depressive Episode With Antidepressant Medication Alone or in Combination With Cognitive Behavioral Therapy: Phase 2 of a 2-Phase Randomized Clinical Trial. JAMA Psychiatry. 2020 Mar 1;77(3):237-245. doi: 10.1001/jamapsychiatry.2019.3900. PMID 31799993
- [Derived] Hollon SD, DeRubeis RJ, Fawcett J, Amsterdam JD, Shelton RC, Zajecka J, Young PR, Gallop R. Effect of cognitive therapy with antidepressant medications vs antidepressants alone on the rate of recovery in major depressive disorder: a randomized clinical trial. JAMA Psychiatry. 2014 Oct;71(10):1157-64. doi: 10.1001/jamapsychiatry.2014.1054. PMID 25142196 (Retraction: PMID 27097060 JAMA Psychiatry. 2016 Jun 1;73(6):639-40)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment into the study started in October 2002 and the last of the 452 patients randomized completed up to three years of treatment and a subsequent three your maintenance/follow-up in July 2012
Groups:
- Cognitive Therapy Plus Antidepressant Medications: Participants will receive antidepressant medication plus cognitive therapy
  Cognitive Therapy (CT): CT sessions occur weekly during acute treatment and monthly during continuation. Acute treatment may last up to 19 months. Remitted patients are continued on medication for up to 42 months from initial randomization until they meet criteria for recovery. At recovery, patients receiving combined treatment discontinue CT.
  Antidepressant medications: Antidepressant medication is distributed as clinically indicated with augmentation and ancillary medications as needed. Acute treatment may last up to 19 months. Remitted patients are continued on medication for up to 42 months from the point of initial randomization until they meet criteria for recovery. All recovered patients are randomized a second time to either maintenance medication or medication withdrawal. Patients are then monitored over 36 months to ascertain risk for recurrence of depressive symptoms.
- Antidepressant Medications Alone: Participants will receive maintenance of antidepressant medication alone
  Antidepressant medications: Antidepressant medication is distributed as clinically indicated with augmentation and ancillary medications as needed. Acute treatment may last up to 19 months. Remitted patients are continued on medication for up to 42 months from the point of initial randomization until they meet criteria for recovery. All recovered patients are randomized a second time to either maintenance medication or medication withdrawal. Patients are then monitored over 36 months to ascertain risk for recurrence of depressive symptoms.
Period: Overall Study
Arm/Group | Cognitive Therapy Plus Antidepressant Medications | Antidepressant Medications Alone
Started | 227 | 225
Completed | 227 | 225
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants met criteria for Major Depressive Disorder (MDD) with exclusions only for psychosis and selected personality disorders
Groups:
- Cognitive Therapy Plus Antidepressant Medications: Participants will receive antidepressant medication plus cognitive therapy
  Cognitive Therapy (CT): CT sessions occur weekly during acute treatment and monthly during continuation. Acute treatment may last up to 18 months. Remitted patients are continued on medication for up to 36 months from initial randomization until they meet criteria for recovery. At recovery, patients receiving combined treatment discontinue CT.
  Antidepressant medications: Antidepressant medication is distributed as clinically indicated with augmentation and ancillary medications as needed. Acute treatment may last up to 18 months. Remitted patients are continued on medication for up to 36 months from the point of initial randomization until they meet criteria for recovery. All recovered patients are randomized a second time to either maintenance medication or medication withdrawal. Patients are then monitored over 36 months to ascertain risk for recurrence of depressive symptoms.
- Antidepressant Medications Alone: Participants will receive maintenance of antidepressant medication alone
  Antidepressant medications: Antidepressant medication is distributed as clinically indicated with augmentation and ancillary medications as needed. Acute treatment may last up to 18 months. Remitted patients are continued on medication for up to 36 months from the point of initial randomization until they meet criteria for recovery. All recovered patients are randomized a second time to either maintenance medication or medication withdrawal. Patients are then monitored over 36 months to ascertain risk for recurrence of depressive symptoms.
- Total: Total of all reporting groups
Arm/Group | Cognitive Therapy Plus Antidepressant Medications | Antidepressant Medications Alone | Total
Number analyzed (Participants) | 227 | 225 | 452
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (12.9) | 43.0 (13.4) | 43.2 (13.1)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 214 | 214 | 428
  >=65 years | 13 | 11 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 136 | 266
  Male | 97 | 89 | 186
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 1 | 5
  Asian | 6 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 21 | 27 | 48
  White | 194 | 193 | 387
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 10 | 27
  Not Hispanic or Latino | 210 | 215 | 425
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 227 | 225 | 452
Number of participants who met criteria for Major Depressive Disorder via SCID-MDD [Number; unit: participants] | 227 | 225 | 452

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Remission According to the Longitudinal Interval Follow-up Evaluation (LIFE) and the Hamilton Rating Scale for Depression (HRSD)
Description: Remission defined as four consecutive weeks of LIFE Problem Symptom Rating (PSR) values of 2 or less and HRSD scores of 8 or less for four consecutive weeks (with partial remission defined as LIFE PSR values of 3 or less and HRSD scores of 12 or less after month 12 only)
Time Frame: Through month 18 of treatment
Measure: Number; unit: number participants that reach remission
Arm/Group | Cognitive Therapy Plus Antidepressant Medications | Antidepressant Medications Alone
Number analyzed (Participants) | 227 | 225
number participants that reach remission | 187 | 170
Statistical Analysis 1: Comparison: Cognitive Therapy Plus Antidepressant Medications vs Antidepressant Medications Alone; Test type: Superiority or Other; p = .038, Subdistribution hazard model

2. Primary Outcome: Number of Participants in Recovery According to the LIFE and HRSD
Description: Six consecutive months following remission without relapse (two weeks of elevated LIFE PSR scores of 4 or more and HRSD scores of 14 and above)
Time Frame: Through 36 months of treatment
Measure: Number; unit: number participants that reach recovery
Groups:
- Antidepressant Medications Only: Participants will receive maintenance of antidepressant medication alone
  Antidepressant medications: Antidepressant medication is distributed as clinically indicated with augmentation and ancillary medications as needed. Acute treatment may last up to 18 months. Remitted patients are continued on medication for up to 36 months from the point of initial randomization until they meet criteria for recovery. All recovered patients are randomized a second time to either maintenance medication or medication withdrawal. Patients are then monitored over 36 months to ascertain risk for recurrence of depressive symptoms.
Arm/Group | Cognitive Therapy Plus Antidepressant Medications | Antidepressant Medications Only
Number analyzed (Participants) | 227 | 225
number participants that reach recovery | 165 | 140
Statistical Analysis 1: Comparison: Cognitive Therapy Plus Antidepressant Medications vs Antidepressant Medications Only; Test type: Superiority or Other; p < 0.01, Subdistribution hazard model

3. Primary Outcome: Number of Participants in Recurrence According to the LIFE and HRSD
Description: Recurrence defined as two consecutive weeks of elevated LIFE PSR scores of 5 or above and HRSD scores of 16 or above (three weeks during period of medication withdrawal)
Time Frame: Measured up to Month 36 from recovery
Measure: Count of Participants; unit: Participants
Groups:
- Prior CBT + Meds Maintained: Patients who recovered on combined treatment (CBT + Meds) were phased out of cognitive therapy and maintained on medications
- Prior CBT + Meds Withdrawn: Patients who recovered on combined treatment (CBT + Meds) were phased out of cognitive therapy and withdrawn from medications
- Prioir Meds Maintained: Patients who recovered on medication treatment were maintained on medications
- Prior Meds Withdrawn: Patients who recovered on medication treatment were withdrawn from medications
Arm/Group | Prior CBT + Meds Maintained | Prior CBT + Meds Withdrawn | Prioir Meds Maintained | Prior Meds Withdrawn
Number analyzed (Participants) | 124 | 103 | 111 | 114
Participants | 78 | 85 | 79 | 103

4. Other Pre Specified Outcome: Serious Adverse Events
Description: Number Serious Adverse Events (SAEs) as reported to the Institutional Review Boards and Data Safety Monitoring Board throughout the duration of the study
Time Frame: Throughout study, up to 54 months
Measure: Number; unit: number of SAE's
Arm/Group | Cognitive Therapy Plus Antidepressant Medications | Antidepressant Medications Only
Number analyzed (Participants) | 227 | 225
number of SAE's | 59 | 82

ADVERSE EVENTS:
Time Frame: Acute treatment up to 18 months and continuation treatment up to 36 months following randomization with subsequent 36 month maintenance phase following recovery
Arm/Group | Cognitive Therapy Plus Antidepressant Medications | Antidepressant Medications Alone
Serious Adverse Events (participants affected / at risk) | 59/227 | 82/225
Other Adverse Events (participants affected / at risk) | 0/227 | 0/225
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Therapy Plus Antidepressant Medications (N=227) | Antidepressant Medications Alone (N=225)
Death (any cause) (General disorders) | 3 (3) | 1 (1)
Suicide Attempt (Psychiatric disorders) | 4 (5) | 8 (9)
Psychiatric Hospitalizations (Psychiatric disorders) | 15 (19) | 28 (36)
Medical Hospitalizations (General disorders) | 30 (46) | 37 (61)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 4 (5) | 5 (6)
Motor Vehicle Accidents (MVA) (General disorders) | 1 (1) | 3 (3)
Other (General disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No